CLINICAL TRIAL: NCT07335003
Title: Prospective Randomized Controlled Study of the Photoprotection and Prevention of Actinic Damage With Anthelios Fluide 100 KA+ UVMune 400 in Patients With Multiple Actinic Keratoses
Brief Title: Study of the Photoprotection and Prevention of Actinic Damage With Anthelios Fluide 100 KA+ UVMune 400 in Patients With Multiple Actinic Keratoses
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cosmetique Active International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: X24-0147 / LRP23028
Record Dates: First submitted 2025-07-04; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Actinic Keratosis (AK)
Keywords: Prevention; Photoprotection; actinic keratosis; diagnosis
MeSH Terms: conditions — Keratosis, Actinic; Disease | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sunscreen investigational product (Active Comparator): Participants (40) will be asked to follow usual recommendations for AK patients as per sun protection information guidelines document provided by Melanoma Institute Australia and will use the sunscreen investigational product at least once every morning and to reapply as often as necessary during the day in case of sun exposure.
  Interventions: Other: Tested product group
- Control Group (Placebo Comparator): Participants (40) will be asked to follow usual recommendations for AK patients as per sun protection information guidelines document provided by Melanoma Institute Australia and may use their normal sun cream
  Interventions: Other: Control group

INTERVENTIONS:
Other: Tested product group — The investigational sunscreen will be applied at least once every morning. Product will be re-applied every 2 hours in case of prolonged exposure or when the likelihood of sunscreen having been removed is high, such as after sweating, water immersion, friction from clothing and exfoliation from sand.
  The investigational product should be applied on all exposed areas. Scalp, face (avoiding eye contours), neck, forearms, back of the hands, and décolleté will be treated every day . The recommended application dose is 2 mg/cm².
  Arms: Sunscreen investigational product
Other: Control group — Participants will be allowed to use the preferred sunscreen (a broad spectrum sunscreen with an SPF of at least 50+) as per their usual routine (every 2 hours and after swimming or exercice).
  Arms: Control Group

SUMMARY:
Participants will be invited to take part in a research study as they have been diagnosed with multiple actinic keratosis lesions (AK). AK usually present as small, rough, dry, scaly and/or crusty patches or papules of the skin that can be skin-coloured pink, red, tan or a combinationof colours and are often easier to feel than see at their earlier stages. AK are commonly diagnosed in adults, particularly in patients aged 45 years and older and are considered to be pre-cancerous lesions.

The research is aiming to investigate the protective effect of an investigational sunscreen known as Anthelios Fluide 100 KA+ UVMune 400, when used together with good sun protection habits (which include staying in the shade during the hours of 11 am and 3 pm, wearing sun-protective clothing, wearing a wide-brimmed hat) in participants with multiple Actinic keratoses's.

Eligible participants will be randomly assigned into 1 of 2 groups - an intervention or control group The study main objective is to evaluate tested sunscreen prevention on actinic keratosis lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Adult outpatients ≥ 60y old with at least 11 clinically typical actinic keratosis lesions, including at least one on the face;
2. Patient having understood and signed a written informed Consent Form to participate in the study indicating the potential participant's willingness to undergo the study procedures and complete the study.

Exclusion Criteria:

1. Atypical actinic keratosis lesions including suspected squamous cell carcinoma and basal cell carcinoma (could be present at screening and treated but cannot be present at 1st visit);
2. History of >2 squamous cell carcinomas;
3. Known history of immunodepression whatever its cause in the past year;
4. Participants who cannot undergo skin biopsies, with a history of scarring problems or who have developed adverse effects from the use of local anesthesia will also be excluded.
5. Participant using interferon or interferon inducers, immunomodulators, cytotoxic or immunosuppressive drugs, corticosteroids, retinoids, other keratolytics or have received investigational drug within 4 weeks before enrolment
6. Participant having active, localized or systemic infection other than the AK lesions
7. Participant having any dermatological affection within the treated and adjacent area according to the Investigator judgement
8. Participant having a present or past skin condition that according to Investigator judgment, deems inappropriate for study participation
9. Participant having other significant medical conditions that according to Investigator Judgment, deems inappropriate for study participation
10. Participant having a known hypersensitivity, allergy or contraindication to any ingredients contained within the cosmetic products,
11. Participant taking part or intending to take part in another study for 30 days prior to D1 visit, and 30 days following last study visit. that according to Investigator judgment, deems inappropriate or may interfere for study participation
12. Participant using light-based devices such as but not limited to PUVA (Psoralen Ultraviolet A therapy), IPL (Intense Pulsed Light), laser, LED (Light Emitting Diode) devices or tanning beds, within 4 weeks before enrolment.
13. Participant having applied any topical product on the investigational areas the day of enrolment visit,
14. Participant under legal guardianship or incapacitation.
15. Participant being psychologically incapable of signing informed Consent Form and unable to comply with the protocol requirements according to investigator judgment.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2029-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
The full body number of Actinic Keratosis lesions | at baseline, 3, 6 and 9 months post commencement of intervention
  Actinic Keratosis clinical evaluation (total number of lesions and severity and location will be recorded)

SECONDARY OUTCOMES:
Variation of the photoprotection index (SEPI) - questionnaire | at baseline, 3, 6 and 9 months post commencement of intervention
  Scoring instrument for assessments of sun habits and sun protection behaviour. It consists of 2 parts: part I addressing the present behaviour and part II addressing propensity to increase sun protection based on the Transtheorical Model of Behaviour Change.
Variation of layers' thickness on Actinic Keratosis lesions | at baseline, 3, 6 and 9 months post-commencement of intervention
  Line-Field Optical Coherence Tomography (LC-OCT) images will be acquired on 2 Actinic Keratosis lesions.
  Measured metric: Thickness of layers (in µm)
Variation of biomarkers of disease severity (p53) | at baseline and 6 months post-commencement of intervention
  using skin biopsy (for morphology, immunohistochemistry) in a subset of participants (10 patients per group)
Questionnaire (self-assessment) | 6 months post-commencement of intervention
  Questions on cosmeticity, efficacy and tolerability of the investigational product tested will be completed by patients. 5 different responses will be proposed (Disagree, Disagree partly, Neither agree neither disagree, Agree and Fully agree)
Adverse Events reporting | at 1, 2, 3, 6 and 9 months post-commencement of intervention
  Any untoward medical occurrence, unintended disease or injury or any untoward clinical signs in patients, users or other persons whether or not related to the investigational product or procedures.
Variation of protusion on Actinic Keratosis lesions | at baseline, 3, 6 and 9 months post-commencement of intervention
  Line-Field Optical Coherence Tomography (LC-OCT) images will be acquired on 2 Actinic Keratosis lesions.
  Measured metric: Protrusion score (grade 1, 2 and 3)
Variation of DEJ undulation on Actinic Keratosis lesions | at baseline, 3, 6 and 9 months post-commencement of intervention
  Line-Field Optical Coherence Tomography (LC-OCT) images will be acquired on 2 Actinic Keratosis lesions.
  Measured metric: Dermal-Epidermal Junction undulation score (in %)
Variation of Keratinocyte nucleus atypia on Actinic Keratosis lesions | at baseline, 3, 6 and 9 months post-commencement of intervention
  Line-Field Optical Coherence Tomography (LC-OCT) images will be acquired on 2 Actinic Keratosis lesions.
  Measured metric: Keratinocyte nucleus atypia score (value between 0 and 1)
Variation of Keratinocyte nucleus morphological characterization on Actinic Keratosis lesions | at baseline, 3, 6 and 9 months post-commencement of intervention
  Line-Field Optical Coherence Tomography (LC-OCT) images will be acquired on 2 Actinic Keratosis lesions.
  Measured metric: morphological characterization (volume, compactness)
Variation of Keratinocyte nucleus distribution on Actinic Keratosis lesions | at baseline, 3, 6 and 9 months post-commencement of intervention
  Line-Field Optical Coherence Tomography (LC-OCT) images will be acquired on 2 Actinic Keratosis lesions.
  Measured metric: Keratinocyte nucleus distribution (density, distribution by layer)

CONTACTS AND LOCATIONS:
Locations (1):
- Sydney Melanoma Diagnostic Centre, Royal Prince Alfred Hospital, Camperdown, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Undecided